CLINICAL TRIAL: NCT00602095
Title: A Randomised Comparison Between Intravaginal Dinoprostone Intravaginal Misoprostol and Transcervical Balloon Catheter for Labour Induction
Brief Title: Labour Induction With Misoprostol, Dinoprostone and Bard Catheter
Acronym: LI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Lena Marions MD PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMS2007; KS2007
Record Dates: First submitted 2008-01-02; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Pregnancy
Keywords: Labor induction; cervical ripening; misoprostol; dinoprostone; balloon catheter; prostaglandin
MeSH Terms: interventions — Misoprostol; Tablets; Dinoprostone; dinoprost tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Labour induction with misoprostol
  Interventions: Drug: misoprostol
- 2 (Active Comparator): Labour induction with dinoprostone
  Interventions: Drug: dinoprostone
- 3 (Experimental): Labour induction with bard
  Interventions: Device: Bard Catheter (balloon catheter)

INTERVENTIONS:
Drug: misoprostol — 0.025mg tablet vaginally every 4 hour until progress
  Other Names: Cytotec, one quarter of a 0.100mg tablet
  Arms: 1
Drug: dinoprostone — 2mg vaginal gel every 6 hours until progress
  Other Names: Minprostin
  Arms: 2
Device: Bard Catheter (balloon catheter) — Intracervical balloon catheter positioned above internal cervical os and filled with sterile water. Removed when cervix was dilated
  Other Names: Bard Catheter
  Arms: 3

SUMMARY:
This is a randomised study aimed at comparing the currently most frequently used prostaglandin dinoprostone to two other methods, the cheaper and perhaps more effective prostaglandin misoprostol and a transcervical catheter. 592 women were recruited and randomised to one of the three methods. The main outcome measures were time to delivery, rate of instrumental deliveries and maternal neonatal outcome. Our hypothesis was that misoprostol would be superior to the other methods.

The main finding of our trial was that the catheter showed the shortest induction to delivery interval. There were no differences between the two other prostaglandins. No differences in maternal and neonatal outcome was found

ELIGIBILITY:
Inclusion Criteria:

* Full term singleton pregnancy with vertex presentation and with an indication for labour induction.
* Absence of active labour
* Bishop score ≤ 6.
* Normal CTG registration

Exclusion Criteria:

* Previous cesarean section
* signs of infection
* immediate need for delivery
* any contraindication for vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2004-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time from treatment start to delivery | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lena Marions, MD PhD, Principal Investigator — Karolinska University Hospital Institute

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264